CLINICAL TRIAL: NCT01988779
Title: Oral Versus Topical Antibiotic Therapy for Treatment of Chronic Rhinosinusitis Exacerbations
Brief Title: Oral Versus Topical Antibiotics for Chronic Rhinosinusitis Exacerbations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Li-Xing Man, M.D., University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 45566
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Chronic Rhinosinusitis
MeSH Terms: interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral placebo with nebulized intranasal levofloxacin (Active Comparator): Placebo oral tablet by mouth daily for 14 consecutive days along with nebulized levofloxacin 125 mg twice daily for 14 consecutive days
  Interventions: Drug: oral levofloxacin; Drug: nebulized levofloxacin
- oral antibiotics with nebulized intranasal placebo (Active Comparator): Levofloxacin 500 mg by mouth once daily for 14 consecutive days, along with intranasal placebo solution twice daily for 14 consecutive days.
  Interventions: Drug: oral levofloxacin; Drug: nebulized levofloxacin

INTERVENTIONS:
Drug: oral levofloxacin
Drug: nebulized levofloxacin

SUMMARY:
The purpose of this study is to treat patients with a diagnosis of chronic rhinosinusitis (CRS) and a history of bilateral endoscopic sinus surgery during times of worsening symptoms and signs of acute infection on nasal endoscopy with one of two treatments: (1) oral antibiotics and twice daily intranasal saline irrigations or (2) oral placebo and twice daily intranasal antibiotic irrigations. The two treatments will be compared to see if there is any difference in patient outcomes. This will help guide treatment strategies for patients with CRS in the future.

DETAILED DESCRIPTION:
See brief summary.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18).
2. Diagnosis of CRS.
3. Worsening sinonasal symptoms.
4. Previous bilateral endoscopic sinus surgery (ESS) (including maxillary antrostomy and anterior ethmoidectomy).
5. English speaking.
6. Open sinuses (open middle meatus bilaterally; determined on endoscopy).
7. Positive sinonasal culture (1+ or greater) with sensitivity to one of the pre-chosen antibiotic regimens.

Exclusion Criteria:

1. Patients < 18 years of age.
2. Treatment with systemic or topical antibiotics within the last 1 month.
3. Pregnant women.
4. Non-English speaking persons.
5. Systemically ill at initial visit necessitating treatment prior to culture data.
6. Allergies to chosen susceptible antibiotics.
7. Sinonasal culture with less than 1+ growth.
8. Multiple organisms grown on culture that are not sensitive to a single antibiotic.
9. Patients with ciliary function disorders (cystic fibrosis, Kartagener's syndrome, ciliary dyskinesia).
10. Patients with immunodeficiencies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Xing Man, MD, MPA, Msc, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Department of Otolaryngology Head and Neck Surgery, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 participants screen failed before randomization to the intervention.
Groups:
- Oral Placebo With Nebulized Intranasal Levofloxacin: Placebo oral tablet by mouth daily for 14 consecutive days along with nebulized levofloxacin 125 mg twice daily for 14 consecutive days
  oral levofloxacin
  nebulized levofloxacin
- Oral Antibiotics With Nebulized Intranasal Placebo: Levofloxacin 500 mg by mouth once daily for 14 consecutive days, along with intranasal placebo solution twice daily for 14 consecutive days.
  oral levofloxacin
  nebulized levofloxacin
Period: Overall Study
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo
Started | 12 | 13
Completed | 9 | 11
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Rhinosinusitis Disability Index (RSDI) Score
Description: The Rhinosinusitis Disability Index is a 30-item questionnaire completed by the patient or subject. Each item has a value of zero to four, a higher score indicates a self-perception of worse symptoms. The minimum score is zero and the maximum score is 120.
  The difference score here is the post-treatment score minus the pre-treatment score, with lower meaning more improvement
Time Frame: Baseline and 14 days after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo
Number analyzed (Participants) | 9 | 11
units on a scale | -8.000 (29.47) | -14.82 (13.49)
Statistical Analysis 1: Comparison: Oral Placebo With Nebulized Intranasal Levofloxacin vs Oral Antibiotics With Nebulized Intranasal Placebo; Test type: Non-Inferiority — Assuming that the non-inferiority limit of topical therapy is 20% of that for oral therapy; p = 0.505, ANOVA

2. Secondary Outcome: Change in Sino-nasal Outcome Test (SNOT-22) Score
Description: The Sino-nasal outcome test is a 22-item questionnaire completed by the patient or subject. Each item has a value of zero to five, a higher score indicates a self-perception of worse symptoms. The minimum score is zero and the maximum score is 110.
  The difference score here is the post-treatment score minus the pre-treatment score, with lower meaning more improvement
Time Frame: Baseline and 14 days after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo
Number analyzed (Participants) | 9 | 11
units on a scale | -2.333 (33.02) | -18.73 (12.37)

3. Secondary Outcome: Change in Bilateral Endoscopy Findings Using POSE Score
Description: The Perioperative Sinus Endoscopy (POSE) instrument is a specific tool to endoscopically assess the sinus cavities of patients who have undergone endoscopic sinus surgery.
  Each POSE score has a minimum of 0 and a maximum of 16, with a higher score indicating a worse outcome.
  Here, the Left and Right POSE scores are summed and the difference between baseline and the 14 day after treatment is reported.
  The change in bilateral POSE score can in principle be -32 to +32, with increased scores indicating worse outcome and negative scores indicating improvement over the treatment period.
Time Frame: Baseline and 14 days after treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo
Number analyzed (Participants) | 9 | 11
units on a scale | -2.889 (5.442) | -4.545 (2.806)
Statistical Analysis 1: Comparison: Oral Placebo With Nebulized Intranasal Levofloxacin vs Oral Antibiotics With Nebulized Intranasal Placebo; Test type: Non-Inferiority — Assuming that the non-inferiority limit of topical therapy is 20% of that for oral therapy; p = 0.390, ANOVA

4. Secondary Outcome: Number of Participants With Post-treatment Culture Negativity
Description: Post-treatment culture negativity, defined as less than 1+ growth of organisms. A subject is counted '1' if both nares are free of bacterial growth, and '0' if growth is 1+ of more
Time Frame: 14 days after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo
Number analyzed (Participants) | 9 | 11
Participants | 5 | 2
Statistical Analysis 1: Comparison: Oral Placebo With Nebulized Intranasal Levofloxacin vs Oral Antibiotics With Nebulized Intranasal Placebo; Test type: Non-Inferiority — Assuming that the non-inferiority limit of topical therapy is 20% of that for oral therapy; p = 0.036, ANOVA

5. Secondary Outcome: Mean Change in the Total Bacterial Community
Description: The bacterial community was determined using a 16S rRNA quantitative PCR processed using Quantitative Insights into Microbial Ecology (QIIME) software, version 1.8 to yield the number of operational taxonomic units in each subject sample. The count has a minimum of zero with an increasing score indicating a larger number of distinct bacterial species.
Time Frame: Baseline and 14 days after treatment
Population: Data was only collected on the first consecutive 8 randomized participants and had equal numbers in each group
Measure: Mean (Standard Deviation); unit: operational taxonomic units
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo
Number analyzed (Participants) | 4 | 4
operational taxonomic units | 17.40 (9.530) | 6.700 (7.404)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Oral Placebo With Nebulized Intranasal Levofloxacin | Oral Antibiotics With Nebulized Intranasal Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 5/12 | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Placebo With Nebulized Intranasal Levofloxacin (N=12) | Oral Antibiotics With Nebulized Intranasal Placebo (N=13)
epistaxis (General disorders) | 3 | 6
Fever (General disorders) | 2 | 0
diarrhea (Gastrointestinal disorders) | 1 | 3
joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
bad taste (Gastrointestinal disorders) | 3 | 3
nausea/vomiting (Gastrointestinal disorders) | 1 | 1
dizziness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT01988779/Prot_SAP_000.pdf